CLINICAL TRIAL: NCT02505347
Title: Early Functional Return to Work Following Distal Biceps Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00057067
Record Dates: First submitted 2015-06-30; First posted 2015-07-22 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2021-09

CONDITIONS: Biceps Tendon Rupture
MeSH Terms: interventions — Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No splint (Experimental): will be able to move the arm as tolerated following surgery.
  Interventions: Other: No splint
- Splint (Active Comparator): will receive a splint following surgery for 6 weeks.
  Interventions: Device: Splint

INTERVENTIONS:
Other: No splint — Can move arm as tolerated with no restrictions on mobility
  Arms: No splint
Device: Splint — Wear splint for 6 weeks, only to remove for rehab and personal care
  Arms: Splint

SUMMARY:
Distal biceps ruptures occur most commonly among young males in their third and fourth decade of life. These injuries are becoming more common, however, as the aging population is remaining active through sport or labour demands. Distal biceps tears or ruptures follow a heavy eccentric load being placed on a shortened or flexed muscle, and often require surgical repair. Functionally, distal biceps injuries cause impairment as this portion of the muscle is largely responsible for supination and flexion at the elbow. Currently there is no consensus regarding post-operative immobilization protocols, and little evidence is available regarding timeframe for early return to functional activities. Existing evidence on functional outcomes post distal biceps tendon repair (DBTR) is of low quality with small sample sizes, and no known RCTs exist comparing early mobilization to immobilization on functional return. Reported timeframes for immobilization range from early controlled motion on day 1 post-operatively to complete immobilization for 6 weeks.

The primary study goal is to determine the effect of immobilization compared to unrestricted mobility post DBTR on early functional return to activities. It has been previously reported that those with DBTR related to a workers compensation injury returned to full duties in 3.95 months, while those with a non-workers compensation related injury returned to full work duties in 1.35 months. In Alberta, near 100 WCB claims were made for DBTR in both 2013 and 2014. Early mobilization of these repairs may allow an earlier return to modified and full work duties, thereby improving the functional quality of life of the individual as well as reducing the overall cost of disability payments.

This study will assess the 1) time to return to pre-injury work level and 2) time to return to modified duties among those who have no movement restriction post-repair and those who are splinted for 6 weeks. Re-rupture rates between groups will also be assessed as will strength, range of motion (ROM) and quality of life. These findings will assist in developing a standardized protocol for immobilization to optimize functional and clinical outcomes while expediting return to work.

DETAILED DESCRIPTION:
Research Questions:

In patients who are immobilized for 6 weeks and those who are allowed unrestricted movement following DBTR, Are there differences during the first post-operative year in:

1. Time to return to work (modified and pre-injury levels)?
2. The proportion of subjects (if any) who re-rupture

a. Strength (flexion, supination) of the elbow b. ROM (flexion, supination) of the elbow c. Self-reported functional quality of life d. Pain between groups

Research Hypotheses:

1. A shorter time to return to work (modified and pre-injury levels) will be identified for the unrestricted movement group compared to the immobilized group.
2. Less than 2% of patients in either group will re-rupture during the first post-operative year.
3. Patients in the unrestricted movement group will have greater early improvements in a) strength; b) ROM; c) functional quality of life scores; and d) pain in the first 3-6 postoperative months compared to those in the immobilized group.

Theoretical significance and practical importance Currently there is no consensus regarding post-operative immobilization protocols, and little evidence is available regarding timeframe for early return to functional activities following DBTR. Existing evidence on functional outcomes post DBTR is of low quality with small sample sizes, and no known RCTs exist comparing early mobilization to immobilization on functional return. Reported timeframes for immobilization range from early controlled motion on day 1 post-operatively to complete immobilization for 6 weeks.

The primary study goal is to determine the effect of immobilization for 6 weeks post-operatively compared to unrestricted mobility post DBTR on early functional return to activities. It has been previously reported that those with DBTR related to a workers compensation injury returned to full duties in 3.95 months, while those with a non-workers compensation related injury returned to full work duties in 1.35 months. In Alberta, near 100 WCB claims were made annually for DBTR in both 2013 and 2014. Early mobilization of these repairs may allow an earlier return to modified and full work duties, thereby improving the functional quality of life of the individual as well as reducing the overall cost of disability payments.

Research plan and methodology Design/Setting: This study is a parallel randomized control trial with computer generated randomization blocks stratified by surgeon. Patient enrollment and follow-up will occur primarily at Sturgeon Community Hospital (SCH).

Sample Size To ensure that the study is properly powered to detect a difference between groups with a power = 0.90, α = 0.05, µ1 = 14 (unrestricted mobility), µ2 = 21 (immobilized), δ = 10, a total of 88 participants is required (44 to each group). To allow for attrition of sample size in the first year, we will enroll up to 100 subjects (50 in each study arm).

This calculation is based on a conservative estimate of a 1 week difference in return to work between groups. If the group differences is greater than 1 week we will remain well-powered. If the group difference is less than 1 week, this is likely not a clinically important difference between groups.

This sample size of 100 should also be sufficient to allow for further sub-analyses between participants who are WCB claimants and those who are not and is adequately powered to compare the secondary and tertiary outcomes between groups, with the exception of re-ruptures, which is expected to be very low in both groups.

Screening and Enrollment Patients will be screened for study eligibility at their initial preoperative clinic visit by the attending surgeon and research coordinator. The research coordinator will track reasons for exclusion, either by patient refusal or surgeon exclusion based on patient characteristics. Those who consent will sign and complete an informed consent form and undergo a baseline evaluation.

Baseline Evaluation: Consented subjects will undergo a pre-operative assessment by a study therapist who is independent of their clinical care. The assessment will consist of 1) baseline demographics form (age, mechanism of injury, past and current medical status, work and activity demands; dominant hand), 2) work-related questions (i.e. occupation, employment status, type of work performed) 3) the Quick Disabilities of the Arm, Shoulder, and Hand questionnaire (Q-DASH), 4) visual analogue scale (VAS) for pain at rest and with activity 5) bilateral elbow ROM in the planes of supination and flexion, 6) bilateral elbow strength for flexion and supination using a handheld dynamometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT), and 7) an ultrasound or MRI to confirm the diagnosis. Imaging at this pre-operative stage is standard of care, and not dependent on study involvement. All data will be collected using standardized forms and entered into a password-protected database.

Intervention

Based upon the surgeons' ability to perform a tension free repair, subjects will be randomized following surgery to either:

1. immobilized for 6 weeks postoperative or
2. unrestricted mobility Those in the immobilized group will be splinted as per current care for 6 weeks, and will remove the splint only for personal care or active-assisted ROM and gentle stretching exercises, as prescribed by an occupational/physical therapist.

Those with unrestricted mobility will be able to move the joint as tolerated post-operatively, but will avoid heavy lifting (>5 pounds) in the first six postoperative weeks.

Those patients who consent, but are excluded at time of surgery will be noted to determine the proportion of patients who are able to participate in an early mobilization regimen. Reasons for exclusion will be recorded.

Rehabilitation Each patient will be referred for a course of physiotherapy post-operatively. Although principles of tissue healing will be followed for both groups, patients in the unrestricted mobility group are likely to start progressive resisted activities by 6-8 weeks post-operatively while the immobilized group will likely not start progressive resisted activities until 8-10 weeks post-operatively. Time (days) of splinting in the immobilized group will be recorded as the time from when the splint was applied post-operatively to the date the splint was fully discontinued. Start and end dates for physiotherapy will be recorded as will the timing of commencing resisted activities.

Follow-up Evaluation Participants will be reassessed by the research coordinator and surgeon at their usual clinic follow-ups at 6 weeks, and 3 and 6 months. Participants will be reassessed by the research coordinator only at 12 months post-operatively.

At each visit outcomes to be recorded will include: current working status (not yet working, modified, full duties) and date of return to any work, ROM measurements, Q-DASH questionnaire, and VAS pain scale. Any complications related to their injury or causing a delay in return to work will also be noted.

Commencing at the 3 month visit and continuing for all subsequent visits, strength will also be assessed using a myometer. Start and end dates of physiotherapy treatment will be recorded to compare the rehabilitation course between groups. Ultrasound imaging will be performed at 12 months, or if there is any history of re-injury to confirm the integrity of the repair.

Analysis We will be using quantitative analytical methods. Descriptive statistics (frequencies, proportions, means and variation) will be determined for all variables.

For the primary outcome (time [days] for return to modified duties) we will use an unpaired t-test to assess for differences between both groups. T-tests will also be used to analyze secondary outcomes (time to return to pre-injury level of work, re-rupture rates, and Q-DASH scores), and time (days) of splinting in the immobilized group will be reported descriptively (mean). Tertiary outcomes (strength, ROM, Q-DASH) will be analyzed using a two-way repeated measure ANOVA to examine the trajectory of recovery between groups.

A further sub-analysis will be performed to assess primary and secondary outcomes between immobilized and unrestricted mobility groups for those who are identified as work related injury compared to non-work related injury using an analysis of covariance (ANCOVA).

All analyses will be two-tailed with a level of significance of α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* male subjects between 18 and 65 years of age
* patient has had a DBTR amenable to surgical repair
* surgeon must be able to obtain a tension-free repair using an endobutton.
* participants must have been working prior to the injury
* patient must be expected to return to work post-injury

Exclusion Criteria:

* females
* outside of the specified age range
* patient with an identified congenital abnormality at the insertion of the distal biceps tendon
* those who have previously ruptured the tendon or those with tendon ruptures resulting from a multi-trauma
* patients with psychiatric illness, cognitive impairment, or health conditions that preclude informed consent
* patients with life expectancy of less than 2 years
* patients who do not speak/read/understand English
* patients with no fixed address or contact information
* patients who are unwilling to complete follow-ups

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Time (days) to return to work on modified duties | 1 year
  Self reported

SECONDARY OUTCOMES:
Time (days) to return to pre-injury level of work | 12 months
  Self reported
Re-rupture rate | 12 months
  Measured by ultrasound at final visit

OTHER OUTCOMES:
Range of Motion | Baseline, 6 weeks, 3 months, 6 months, 12 months
  Using standard goniometry.
Elbow strength (flexion, supination) | baseline, 6 weeks, 3 months, 6 months, 12 months
  Using myometer. Measured bilaterally at baseline visit.
Quick - DASH | baseline, 6 weeks, 3 months, 6 months, 12 months
Pain VAS | baseline, 6 weeks, 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Beaupre, PT, PhD, Principal Investigator — University of Alberta
Locations (1):
- Sturgeon Community Hospital, St. Albert, Alberta, Canada

REFERENCES:
- [Background] Bergman JW, Silveira A, Chan R, Lapner M, Hildebrand KA, Le ILD, Sheps DM, Beaupre LA, Lalani A. Is Immobilization Necessary for Early Return to Work Following Distal Biceps Repair Using a Cortical Button Technique?: A Randomized Controlled Trial. J Bone Joint Surg Am. 2021 Oct 6;103(19):1763-1771. doi: 10.2106/JBJS.20.02047. PMID 34166263
- See also: Study Video Summary — https://www.youtube.com/watch?v=M5qLlTl69gg
- See also: OrthoEvidence — https://myorthoevidence.com/AceReports/Report/14139?token=98ca3a45-2c20-474d-b147-3a8a27b79880